CLINICAL TRIAL: NCT01075763
Title: Pilot Trial of Interferon Beta-1a in Alzheimer's Disease
Brief Title: A Pilot Trial of Interferon Beta-1a in Alzheimer's Disease
Acronym: REAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.P.A., Italy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24386
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Results first posted 2012-04-04 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's; Dementia; Interferon beta-1a; Rebif
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Interferon beta-1a

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Treatment arm - Rebif® (Experimental): Subjets in this arm received interferon beta-1a (Rebif® 22 mcg tiw)
  Interventions: Drug: Interferon beta-1a
- Placebo arm (Placebo Comparator): Subjects in this arm received placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Interferon beta-1a — Interferon (IFN) beta-1a [Rebif® 22 microgram (mcg), three times per week (tiw)] administered subcutaneously (sc)
  Other Names: Rebif®
  Arms: Treatment arm - Rebif®
Drug: Placebo — The inactive substance (placebo) looks the same as Interferon beta-1a (Rebif®), and is given the same way
  Arms: Placebo arm

SUMMARY:
This was a 52-week, multicentric, phase II, pilot study conducted in 40 subjects with early-onset Alzheimer's disease (AD) to evaluate safety, tolerability and clinical efficacy of subcutaneous (sc) interferon (IFN) beta-1a [Rebif® 22 microgram (mcg), three times per week (tiw)] in the treatment of AD by comparing the neuropsychological performance changes into placebo and treatment arms from screening/baseline to 52 week.

DETAILED DESCRIPTION:
Alzheimer's disease is characterized by progressive cognitive impairment resulting from neuronal loss. The primary pathological feature of the disease is the extracellular deposition of fibrillary amyloid and its compaction into senile plaques. The senile plaque is the focus of a complex cellular reaction involving the activation of both microglia and astrocytes adjacent to the amyloid plaque. In fact, microglias are the most abundant and prominent cellular components associated with these plaques. Plaque-associated microglia exhibits a reactive or activated phenotype. Through the acquisition of a reactive phenotype, microglia responds to various stimuli, as is evident by the increased expression of numerous cell-surface molecules, including major histocompatibility complex (MHC) class-II antigens and complement receptors.

Traditionally, multiple sclerosis (MS) has been considered a "demyelinating" disease. Recent immunocytochemical studies suggest that MS may be more than a demyelinating disorder, and that even in early stages of the disease, MS pathological scenario envisages axonal damage. Interferons, the modern therapeutic strategies for the treatment of MS, are cytokines - proteins which lead to a network of signals within different cells. In the immune system, IFNs act at different levels. For example, IFNs increase the expression of MHC class II antigens and, thereby, facilitate the antigen-presenting process and the activation of lymphocytes. T-lymphocytes are important targets of IFN immunomodulation. In MS, it is believed that IFN beta suppresses the production of proinflammatory cytokines such as IFN-γ and TNF-α, and increases the production of immunosuppressive cytokines such as interleukin-4 (IL-4) and IL-10. Since the activation of microglia and astrocytes is common to both AD and MS, IFN beta could have therapeutic applications in the treatment of AD. Furthermore, recent studies have also found that through astrocyte production, IFNs promote the activation of nerve-growth factor.

OBJECTIVES

* To evaluate safety, tolerability and clinical efficacy of IFN beta-1a (Rebif® 22 mcg, tiw) in the treatment of AD

In this study, subjects were randomized into two groups: the first group (treatment arm, n=20) received Rebif® 22 mcg tiw; the second group (placebo arm, n=20) received placebo. The treatment period was for 28 weeks and subjects were followed up to Week 52. Efficacy was determined by comparing neuropsychological performance changes into placebo and treatment arms from screening/baseline to Week 52.

On Day 1 of the study treatment period, subjects received injection training and were administered the first dose of Rebif under the supervision of the clinical personnel by subcutaneous injection tiw at approximately the same time each day preferably in the late afternoon or evening. All subjects received 28 weeks of therapy and after 24 weeks from the therapy conclusion, a termination visit was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 50 and 75 years
* Subjects diagnosed with AD, according to the Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV)
* Subjects with MMSE score of 20 to 26 (inclusive)
* Subjects supervised by a caregiver
* Subjects who have been given informed written consent and approval of the Local Ethical Committee

Exclusion Criteria:

* Subjects with constant use in the 3 months prior study enrolment of other drugs that can modify the course of the disease (e.g. statins, nonsteroidal anti-inflammatory drugs [NSAIDs] and steroids) or symptomatic cognitive treatments (e.g. cholinesterase inhibitors)
* Subjects with modified Hachinski Ischemic Score ≥ 4
* Subjects who are unable to undergo neuropsychological evaluation (including analphabetism)
* Subjects with significant liver (aspartate aminotransferase, alanine aminotransferase , alkaline phosphatase > 2.0 times the upper limit of normal [ULN] of the local laboratory, or total bilirubin > 1.5 times the ULN of the local laboratory), thyroid (according to clinical judgment) or hematological dysfunctions (e.g. leucocytes ≤ 2.0 * 109/Liter [L]; platelets ≤ 100 * 109/L; hemoglobin ≤ 12 gram/deciliter [g/dL] for women and ≤ 13 g/dL for men, serum albumin ≤ 3 g/dL)
* Subjects with history (past or recurrent) of depression unresponsive to medication or past medical history of suicidal ideation
* Subjects with severe cardiac disease (angina, congestive heart failure class 3-4 New York Heart Association [NYHA] Functional Classification , or severe arrhythmia)
* Subjects with epilepsy
* Subjects with concomitant use of hypnotic, anxiolytic, antidepressant, antipsychotic, anticholinergic
* Subjects with known allergic reactions against IFNs or other components of the applied drug

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Paolillo, MD, PhD, Study Director — Merck Serono S.P.A., Italy
Locations (1):
- U.VA. Neurologia - Azienda Ospedaliera Garibaldi Nesina, Catania, CT, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- Rebif 22 Mcg: Single dose of interferon beta-1a (Rebif) injection administered subcutaneously (sc) three times per week (tiw) at a dose of 4.4 microgram (mcg) for first 2 weeks followed by 11 mcg for next 2 weeks and finally 22 mcg for remaining 24 weeks (treatment period 28 weeks).
- Placebo: Single dose of matching placebo injection administered sc tiw at a dose of 4.4 mcg for first 2 weeks followed by 11 mcg for next 2 weeks and finally 22 mcg for remaining 24 weeks (treatment period of 28 weeks).
Period: Overall Study
Arm/Group | Rebif 22 Mcg | Placebo
Started | 23 | 19
Completed | 19 | 15
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 2 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rebif 22 Mcg | Placebo | Total
Number analyzed (Participants) | 23 | 19 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.00 (9.08) | 64.58 (6.41) | 63.71 (7.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer's Disease Assessment Scale, Cognitive Subscale (ADAS-Cog) Score
Description: ADAS: global rating scale created to evaluate both cognitive and functional aspects linked with disease progression. ADAS-Cog: subscale of ADAS which consists in a series of short tests aimed to evaluate possible cognitive impairment due to disease progression. It includes 11 items, testing word-finding difficulty, following commands, naming: objects and fingers, orientation, word recognition, recall of test instructions, constructions, ideational praxis, spoken language ability, comprehension of spoken language and word recall. Scores range from 0 (no impairment) to 70 (serious deficit).
Time Frame: Baseline and Week 52
Population: Per protocol population included all participants who received treatments as scheduled and were followed up to week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Rebif 22 Mcg: Single dose of interferon beta-1a (Rebif®) injection administered subcutaneously (sc) three times per week (tiw) at a dose of 4.4 microgram (mcg) for first 2 weeks followed by 11 mcg for next 2 weeks and finally 22 mcg for remaining 24 weeks (treatment period 28 weeks).
Arm/Group | Rebif 22 Mcg | Placebo
Number analyzed (Participants) | 19 | 15
units on a scale
  Baseline | 18.63 (7.86) | 19.81 (6.15)
  Week 52 | 20.66 (9.55) | 20.33 (10.05)
Statistical Analysis 1: Comparison: Rebif 22 Mcg vs Placebo; For baseline: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.64, t-test, 2 sided
Statistical Analysis 2: Comparison: Rebif 22 Mcg vs Placebo; For Week 52: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.92, t-test, 2 sided

2. Secondary Outcome: Alzheimer's Disease Assessment Scale, Cognitive Subscale (ADAS-Cog) Score
Description: as for outcome 1
Time Frame: Week 12 and 28
Population: Per protocol population included all participants who received treatments as scheduled and were followed up to week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rebif 22 Mcg | Placebo
Number analyzed (Participants) | 19 | 15
units on a scale
  Week 12 | 16.74 (6.94) | 17.97 (6.28)
  Week 28 | 18.49 (8.72) | 17.55 (7.02)
Statistical Analysis 1: Comparison: Rebif 22 Mcg vs Placebo; For Week 12: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.63, t-test, 2 sided
Statistical Analysis 2: Comparison: Rebif 22 Mcg vs Placebo; For Week 28: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.74, t-test, 2 sided

3. Secondary Outcome: Mini Mental Status Examination (MMSE) Score
Description: MMSE is a tool for screening cognitive decline associated with dementia. It is a brief examination intended to evaluate an adult participant's level of cognitive functioning. The test is performed in following areas: orientation in time and place, learning and immediate recall, mental control and concentration, short-term recall, naming ability, language expression, verbal comprehension, writing comprehension, writing ability and visual-spatial coordination. Scores range between 0 (maximum cognitive deficit) and 30 (no cognitive deficit).
Time Frame: Baseline, Week 12, 28 and 52
Population: Per protocol population included all participants who received treatments as scheduled and were followed up to week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rebif 22 Mcg | Placebo
Number analyzed (Participants) | 19 | 15
units on a scale
  Baseline | 23.46 (2.14) | 22.93 (1.79)
  Week 12 | 24.50 (3.22) | 24.66 (3.14)
  Week 28 | 24.25 (3.37) | 23.66 (4.92)
  Week 52 | 22.43 (5.33) | 21.98 (5.32)
Statistical Analysis 1: Comparison: Rebif 22 Mcg vs Placebo; For baseline: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.45, t-test, 2 sided
Statistical Analysis 2: Comparison: Rebif 22 Mcg vs Placebo; For Week 12: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.88, t-test, 2 sided
Statistical Analysis 3: Comparison: Rebif 22 Mcg vs Placebo; For Week 28: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.68, t-test, 2 sided
Statistical Analysis 4: Comparison: Rebif 22 Mcg vs Placebo; For Week 52: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.81, t-test, 2 sided

4. Secondary Outcome: Alzheimer's Disease Assessment Scale, Non-cognitive Subscale (ADAS-NonCog) Score
Description: ADAS-NonCog is a subscale of ADAS aimed to evaluate the non-cognitive features such as mood state and behavioral changes. It takes about 10 minutes to be performed and includes 10 items: testing tearful, depressed mood, concentration/distractibility, uncooperative to testing, delusions, hallucinations, pacing, motor activity increase, tremors and appetite change. Scores range between 0 (excellent performance) and 35 (worst performance).
Time Frame: Baseline, Week 12, 28 and 52
Population: Per protocol population included all participants who received treatments as scheduled and were followed up to week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rebif 22 Mcg | Placebo
Number analyzed (Participants) | 19 | 15
units on a scale
  Baseline | 4.37 (4.13) | 6.07 (5.01)
  Week 12 | 3.53 (3.24) | 4.73 (4.27)
  Week 28 | 4.63 (4.36) | 5.20 (3.43)
  Week 52 | 5.47 (5.17) | 7.20 (6.97)
Statistical Analysis 1: Comparison: Rebif 22 Mcg vs Placebo; For baseline: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.29, t-test, 2 sided
Statistical Analysis 2: Comparison: Rebif 22 Mcg vs Placebo; For Week 12: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.36, t-test, 2 sided
Statistical Analysis 3: Comparison: Rebif 22 Mcg vs Placebo; For Week 28: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.68, t-test, 2 sided
Statistical Analysis 4: Comparison: Rebif 22 Mcg vs Placebo; For Week 52: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.41, t-test, 2 sided

5. Secondary Outcome: Instrumental Activities of Daily Living (IADL) Score
Description: IADL is used to evaluate participants with early-stage disease, both to assess level of disease and to determine participant's ability of self-care. IADL scale measures functional impact of emotional, cognitive, and physical impairments. It provides information about participants' compromising rate and care he might need. It includes 8 items: testing ability to use telephone, shopping, food preparation, housekeeping, laundry, mode of transportation, responsibility for own medication and ability to handle finances. Scores range between 0 (impairment) and 8 (full independence).
Time Frame: Baseline, Week 28 and 52
Population: Per protocol population included all participants who received treatments as scheduled and were followed up to week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rebif 22 Mcg | Placebo
Number analyzed (Participants) | 19 | 15
units on a scale
  Baseline | 6.11 (1.45) | 6.20 (1.57)
  Week 28 | 5.84 (1.17) | 5.60 (1.68)
  Week 52 | 4.89 (1.85) | 5.67 (1.63)
Statistical Analysis 1: Comparison: Rebif 22 Mcg vs Placebo; For baseline: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.86, t-test, 2 sided
Statistical Analysis 2: Comparison: Rebif 22 Mcg vs Placebo; For Week 28: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.62, t-test, 2 sided
Statistical Analysis 3: Comparison: Rebif 22 Mcg vs Placebo; For Week 52: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.21, t-test, 2 sided

6. Secondary Outcome: Physical Self-Maintenance Scale (PSMS) Score
Description: PSMS designed as a disability measure for use in planning and evaluating treatment in elderly participants living in community or in institutions, is Guttman scale containing 6 items of self-care. The scale is based on theory that human behavior can be ordered in a hierarchy of complexity, within each category, a further hierarchy of complexity runs from basic to complex activities. It includes 6 items, testing the following areas: toilet use, eating, dressing, physical appearance, deambulation and bath. Scores range between 0 (excellent performance) and 30 (worst performance).
Time Frame: Baseline, Week 28 and 52
Population: Per protocol population included all participants who received treatments as scheduled and were followed up to week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rebif 22 Mcg | Placebo
Number analyzed (Participants) | 19 | 15
units on a scale
  Baseline | 6.42 (1.02) | 6.40 (0.91)
  Week 28 | 6.74 (1.37) | 7.00 (2.65)
  Week 52 | 7.79 (3.34) | 6.87 (1.68)
Statistical Analysis 1: Comparison: Rebif 22 Mcg vs Placebo; For baseline: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.95, t-test, 2 sided
Statistical Analysis 2: Comparison: Rebif 22 Mcg vs Placebo; For Week 28: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.73, t-test, 2 sided
Statistical Analysis 3: Comparison: Rebif 22 Mcg vs Placebo; For Week 52: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.30, t-test, 2 sided

7. Secondary Outcome: Clinician's Interview Based Impression of Change (CIBIC-PLUS) Score
Description: CIBIC-PLUS: structured instrument based on comprehensive evaluation of 3 domains: participant cognition, behavior and functioning, including assessment of daily living activities. It includes 15 items and represents assessment of skilled clinician using validated scales based on the observation at interviews conducted separately with participant and caregiver familiar with behavior of participant. According to comparison between baseline and follow-up assessments, scores can range between 1 (markedly improved) and 7 (markedly worsened), with 4 indicating no change observed between two visits.
Time Frame: Week 28 and 52
Population: Per protocol population included all participants who received treatments as scheduled and were followed up to week 52.
Measure: Number; unit: participants
Arm/Group | Rebif 22 Mcg | Placebo
Number analyzed (Participants) | 19 | 15
participants
  Week 28: CIBIC-PLUS Score 1 | 1 | 0
  Week 28: CIBIC-PLUS Score 2 | 0 | 2
  Week 28: CIBIC-PLUS Score 3 | 7 | 6
  Week 28: CIBIC-PLUS Score 4 | 8 | 5
  Week 28: CIBIC-PLUS Score 5 | 3 | 0
  Week 28: CIBIC-PLUS Score 6 | 0 | 2
  Week 28: CIBIC-PLUS Score 7 | 0 | 0
  Week 52: CIBIC-PLUS Score 1 | 0 | 0
  Week 52: CIBIC-PLUS Score 2 | 0 | 2
  Week 52: CIBIC-PLUS Score 3 | 6 | 2
  Week 52: CIBIC-PLUS Score 4 | 7 | 4
  Week 52: CIBIC-PLUS Score 5 | 1 | 4
  Week 52: CIBIC-PLUS Score 6 | 4 | 3
  Week 52: CIBIC-PLUS Score 7 | 1 | 0

8. Secondary Outcome: Geriatric Depression Scale (GDS) Score
Description: The GDS consists of 30 'yes' or 'no' items aimed to assess depression. One point is assigned to each answer and the cumulative score is rated on a scoring grid. Scores are grouped as follows: 0-9 'normal', 10-19 'mildly depressed', and 20-30 'severely depressed'.
Time Frame: Baseline, Week 28 and 52
Population: Per protocol population included all participants who received treatments as scheduled and were followed up to week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rebif 22 Mcg | Placebo
Number analyzed (Participants) | 19 | 15
units on a scale
  Baseline | 10.11 (6.13) | 10.67 (6.53)
  Week 28 | 9.68 (5.74) | 9.07 (4.32)
  Week 52 | 10.79 (5.93) | 7.50 (5.56)
Statistical Analysis 1: Comparison: Rebif 22 Mcg vs Placebo; For baseline: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.80, t-test, 2 sided
Statistical Analysis 2: Comparison: Rebif 22 Mcg vs Placebo; For Week 28: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.74, t-test, 2 sided
Statistical Analysis 3: Comparison: Rebif 22 Mcg vs Placebo; For Week 52: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.12, t-test, 2 sided

9. Secondary Outcome: Global Deterioration Scale Score
Description: Global deterioration scale includes seven different diagnostic stages ranging between "no cognitive deterioration" and "very serious cognitive deterioration". It investigates the cognitive impairment. Scores range between 1 (no cognitive deterioration) and 7 (very severe cognitive decline).
Time Frame: Baseline, Week 28 and 52
Population: Per protocol population included all participants who received treatments as scheduled and were followed up to week 52.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rebif 22 Mcg | Placebo
Number analyzed (Participants) | 19 | 15
units on a scale
  Baseline | 3.00 (0.47) | 2.87 (0.74)
  Week 28 | 3.05 (0.78) | 3.00 (0.93)
  Week 52 | 3.26 (0.81) | 3.20 (1.08)
Statistical Analysis 1: Comparison: Rebif 22 Mcg vs Placebo; For baseline: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.53, t-test, 2 sided
Statistical Analysis 2: Comparison: Rebif 22 Mcg vs Placebo; For Week 28: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.85, t-test, 2 sided
Statistical Analysis 3: Comparison: Rebif 22 Mcg vs Placebo; For Week 52: the difference between the two groups was analyzed using t-test; Test type: Superiority or Other; p = 0.85, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Baseline to Week 52
Description: An adverse event (AE) was defined as any untoward medical occurrence in the form of signs, symptoms, abnormal laboratory findings, or diseases that emerges or worsens relative to baseline during a clinical study with an Investigational Medicinal Product (IMP), regardless of causal relationship and even if no IMP has been administered.
Arm/Group | Rebif 22 Mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/19
Other Adverse Events (participants affected / at risk) | 5/23 | 5/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rebif 22 Mcg (N=23) | Placebo (N=19)
Articular Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Fever (General disorders) | 1 | 0
High Cholesterol (Investigations) | 3 | 0
High level of alanine transaminase (ALT) and aspartate aminotransferase (AST) (Investigations) | 1 | 0
High level of aspartate aminotransferase (AST) - alanine transaminase (ALT) (Investigations) | 0 | 1
High pseudocholinesterase (Investigations) | 2 | 1
High triglycerides (Investigations) | 1 | 0
High thyroid stimulating hormone (Investigations) | 0 | 1
Low blood pressure (Vascular disorders) | 0 | 1
Repolarization ventricular anomaly (Investigations) | 1 | 0
Right ear buzzing (Ear and labyrinth disorders) | 0 | 1
Flu-like syndrome (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other